CLINICAL TRIAL: NCT03039725
Title: Vaccination Rates in Obstetric Opioid-Addicted Patients
Brief Title: Vaccination Compliance
Status: Completed | Type: Observational
Sponsor: Jaye Shyken, MD (Other)
Responsible Party: Sponsor-Investigator, Jaye Shyken, MD, Principal Investigator, St. Louis University
Organization: St. Louis University (Other)
Other Study IDs: 27919
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Vaccine Compliance
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Retrospective chart review on vaccine compliance

SUMMARY:
Retrospective study to assess a single Clinic on Immunization Practices (ACIP) recommendations for hepatitis A, hepatitis B, influenza, tetanus/diphtheria/pertussis, HPV and pneumococcal disease

DETAILED DESCRIPTION:
Vaccines are known as one of the greatest public health achievements of the twentieth century. Due to the successful implementation of childhood immunization programs in the United States (US), once common disease states such as polio, smallpox, and measles are no longer a natural part of childhood. Unfortunately, these successes have not been replicated in the adult population despite the availability of vaccines and published recommendations guiding appropriate screening for and administration of vaccines. On average, 42,000 adults compared to 300 children die in the US of vaccine-preventable infections every year. In fact, results of the National Health Interview Survey from 2012 demonstrated low immunization rates for adults 19 years of age and older leaving a significant portion of eligible patients susceptible to disease.

Vaccine administration rates are often lower in the obstetric population likely due to fear of administration during pregnancy and lack of recommendations and education to patients about vaccines. The influenza and Tdap vaccines are recommended for every pregnant patient. However, in 2015-16 influenza season only 49.9% of pregnant patients received the influenza vaccine. Additionally, only 30-53.% have receive the Tdap vaccine. Besides these needed vaccines, patients are often indicated for additional vaccines including hepatitis A, hepatitis B, pneumococcal-23, and human papillomavirus. Additionally, patients who have unequivocal or negative rubella titers during pregnancy should receive the measles, mumps, and rubella vaccine when post-partum. Because of the lack of vaccination, the American College of Obstetricians and Gynecologists (ACOG) has recommended that vaccines become part of the routine obstetric care.

According to American Society of Healthcare Pharmacists (ASHP) Guidelines on the pharmacist's role in immunizations, all pharmacists can contribute to the effort by promoting proper immunizations in various ways. One way is by helping to identify patients in need of immunizations by gathering immunization histories, identifying patient specific indication, issuing immunization records to patients, and educating patients on their specific indications, and the risk of the immunizations.

The investigator's team includes a maternal fetal medicine specialist, nurse practitioners, clinical pharmacist, social workers, and registered nurses. The pharmacist meets with all patients to perform medication reconciliation, vaccine history, social history, allergy history, disease specific review of systems, pregnancy related review of systems, and preventative health review; assess medical and preventative health problems; recommend appropriate management of medical problems and preventative health; and provide extensive education including information on all indicated vaccines. The indicated vaccines are recommended to either the physician or nurse practitioner provider for that visit as well as documented in the medical record. Additionally, prior to each office visit, the pharmacist reviews each patient's chart to determine what vaccines are indicated for this visit. This list of indicated vaccines is provided to the nurse who asks the patients about receiving the vaccine at that day's visit. If the patient is willing to receive the vaccine, the nurse has the provider order the indicated vaccines. All the vaccines are kept as floor stock in the clinic to minimize wait time for the patient.

Although there have been recent efforts to increase immunization rates throughout the health care system, there is little evidence about the impact of pharmacists' involvement on immunization rates in outpatient obstetric clinic setting. The goal of this study is to evaluate immunization administration compliance with the Centers for Disease Control (CDC) 2016 immunization recommendations for influenza, pneumococcal 23 polyvalent, hepatitis A, hepatitis B, tetanus, diphtheria, and acellular pertussis (Tdap), human papillomavirus (HPV), and measles-mumps-rubella (MMR).

ELIGIBILITY:
Inclusion Criteria:

* Patients addicted to opioids during pregnancy

Exclusion Criteria:

* must meet inclusion criteria

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Female
  * All ethnic backgrounds
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
compliance with the 2016 ACIP recommendations | 6 months
  Chart review

CONTACTS AND LOCATIONS:
Overall Officials: Jaye Shyken, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No